CLINICAL TRIAL: NCT04938167
Title: Preductal Oxygen Saturation Target in Term and Late Preterm Neonates With Hypoxemic Respiratory Failure or Pulmonary Hypertension (POST-IT)
Brief Title: Preductal Oxygen Saturation Target in Term and Late Preterm Neonates With Hypoxemic Respiratory Failure or Pulmonary Hypertension
Acronym: POST-IT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1766675; 5KL2TR001859-04 (NIH)
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-05

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn; Hypoxemic Respiratory Failure
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized assignment to Standard arm (target preductal SpO2 91% to 95%) or Intervention arm (target preductal SpO2 95% to 99%)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (No Intervention): target preductal SpO2 - 91 to 95%
- Intervention arm (Experimental): target preductal SpO2 - 95 to 99%
  Interventions: Other: 95% - 99% SpO2 target

INTERVENTIONS:
Other: 95% - 99% SpO2 target — If the infant is randomized to the intervention arm, the oxygen saturation goal will be changed from the standard goal of 91% - 95% to the experimental goal of 95%-99%. The treating medical team will then adjust the oxygen and respiratory support to maintain these goals (SpO2 alarm levels will be set at 93% and 100%).
  Arms: Intervention arm

SUMMARY:
The purpose of this research is to evaluate two oxygen saturation goals for newborns with pulmonary hypertension. Participation in this research will involve random assignment to one of two oxygen saturation goals, review of the medical record and targeted echocardiograms.

DETAILED DESCRIPTION:
Successful transition at birth is dependent on establishment of lungs as the organ of gas exchange. Breathing at birth and an increase in alveolar oxygen tension (PAO2) leads to an 8-10 fold increase in pulmonary blood flow with a marked reduction in pulmonary vascular resistance (PVR). Failure to decrease PVR at birth results in hypoxemic respiratory failure (HRF) and persistent pulmonary hypertension of the newborn (PPHN). Hypoxemia exacerbates PPHN by increasing PVR. However, administration of excess oxygen in animal studies has been shown to increase free radical formation and reduce response to pulmonary vasodilators such as inhaled nitric oxide (iNO).

Thus, there is potential for benefit and also poor outcomes at both higher and lower oxygen saturations (SpO2), with the ideal range being unknown. The investigators will conduct a randomized unblinded, pilot trial to compare two ranges of target preductal SpO2 in late preterm and term infants with HRF or PPHN. During this trial the investigators will assess the reliability of a hypoxic respiratory failure/pulmonary hypertension (HRF/PH) score that could then be used in a larger clinical trial. The investigators will also assess trial feasibility and obtain preliminary estimates of outcomes. Our central hypothesis is that neonates with pulmonary hypertension (PH) and/or HRF, targeting preductal SpO2 of 95-99% (intervention) will result in lower PVR and lower need for non-oxygen based pulmonary vasodilators (iNO, milrinone and sildenafil) compared to a target of 91-95% (standard).

ELIGIBILITY:
Inclusion Criteria:

* Corrected gestational age (postmenstrual age) > 34 6/7 weeks
* postnatal age ≤ 28 d
* on respiratory support with invasive mechanical ventilation, non-invasive ventilation, CPAP or high flow nasal cannula (defined as flow rates ≥ 2 LPM with a humidifier), inspired oxygen concentration, FiO2 ≥ 0.3
* and echocardiography shows any finding suggestive of PH (or score > 0 for PH in table 2).
* Infants with congenital diaphragmatic hernia (CDH), Down syndrome, hypoxic ischemic encephalopathy (HIE) on therapeutic hypothermia and patent ductus arteriosus (PDA), patent foramen ovale/atrial septal defect (PFO/ASD) and ventricular septal defect (VSD) (single or multiple) < 2 mm can be included in the study.

Exclusion Criteria:

* < 32 weeks gestation at birth (31 6/7 or lower)
* Weight < 2000 g at the time of enrollment
* Severe HRF with OI > 35 or SpO2 < 75% on FiO2 = 1.0 on mechanical ventilation for > 60 minutes in spite of correction of reversible factors such as pneumothorax
* A condition or congenital anomaly known to be lethal (high likelihood of death during infancy) - e.g., trisomy 18 or trisomy 13
* Congenital heart disease other than ASD/PFO, PDA or VSD (single or multiple defects) < 2 mm.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hypoxemic Respiratory Failure and Pulmonary Hypertension (HRF/PH) score | At enrollment
  Most randomized trials evaluating PPHN have taken oxygenation, echocardiographic evidence of PH or survival with extracorporeal membrane oxygenation (ECMO) as primary endpoints. Oxygenation was primarily assessed with postductal arterial gases. More recently, preductal SpO2 and blood gases have been shown to have advantages during management of PPHN with congenital diaphragmatic hernia (CDH). Given the low need for ECMO in PPHN (other than due to CDH), the investigators have developed a HRF/PH score combining oxygenation using preductal SpO2 and echocardiographic parameters. The score ranges from 0 to 15, with a higher score corresponding to worse respiratory failure or pulmonary hypertension. The primary aim of this pilot trial to understand the variation of this score at two oxygen saturation targets and assess its reliability and validity.
Correlation of the Oxygenation and Echocardiography components of the HRF/PH scores | At enrollment

SECONDARY OUTCOMES:
Intracluster correlation coefficients of the HRF/PH score | Days 3-7
  The investigators will fit a sequence of two-level multilevel models to estimate intracluster correlation coefficients based on the between-infant (level 2) and other relevant variance component(s), after adjusting for fixed effects, including study arm and sex. Interrater reliability at specific days will be estimated by having two or more raters (level 1) score each infant's underlying oxygenation and echocardiography measurements, while within-infant, over-time intracluster correlation will be estimated by analyzing a data set with one score per infant per day (level 1), with fixed effects added to account for day effects and possibly restricted to a smaller number of the later days (e.g. days 3 to 7), in case early-day values are grossly unstable.
Preliminary estimates of intervention effects on outcomes (length of stay, duration of mechanical ventilation, and ECMO) | Day 7
  For obtaining preliminary estimates of intervention effects on Day-7 HRF/PH, the investigators will use the results of Outcome 1 to inform our choice of how best to account for the baseline HRF/PH score, although the investigators anticipate that the within-infant correlation will be suitably modest that ANCOVA-like approaches will be preferred over differences-in-differences. Intervention effects and other regression-parameters will be estimated with robust 95% confidence intervals, to ensure accurate coverage.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California-Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siefkes H, Sunderji S, Vaughn J, Sankaran D, Vali P, Vadlaputi P, Timberline S, Bhatt A, Tancredi D, Lakshminrusimha S. Factors to Consider to Study Preductal Oxygen Saturation Targets in Neonatal Pulmonary Hypertension. Children (Basel). 2022 Mar 11;9(3):396. doi: 10.3390/children9030396. PMID 35327768
- See also: Learn more or sign up for the study here! — https://studypages.com/s/testing-levels-of-oxygen-in-newborns-with-pulmonary-hypertension-800422/